CLINICAL TRIAL: NCT02858076
Title: Intravitreous Anti-VEGF vs. Prompt Vitrectomy for Vitreous Hemorrhage From Proliferative Diabetic Retinopathy
Brief Title: Anti-VEGF vs. Prompt Vitrectomy for VH From PDR
Acronym: AB
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Regeneron Pharmaceuticals (Industry); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRCR.net Protocol AB; EY14231 (Other Grant/Funding Number: National Eye Institute); EY23207 (Other Grant/Funding Number: National Eye Institute); EY18817 (Other Grant/Funding Number: National Eye Institute)
Record Dates: First submitted 2016-08-03; First posted 2016-08-08 (Estimated); Results first posted 2021-01-19 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-02

CONDITIONS: Proliferative Diabetic Retinopathy; Vitreous Hemorrhage
Keywords: Anti-VEGF; Vitrectomy
MeSH Terms: conditions — Vitreous Hemorrhage | interventions — aflibercept

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravitreous 2 mg aflibercept injections (Active Comparator): Initial injection must be given on the day of randomization. Follow-up injections will be performed as often as every 4 weeks unless criteria for deferral are met.
  Interventions: Drug: 2-mg Intravitreous Aflibercept Injection
- Prompt vitrectomy plus panretinal photocoagulation (Active Comparator): For the prompt vitrectomy + panretinal photocoagulation group, the vitrectomy must be scheduled to be performed within 2 weeks of randomization. Vitrectomy will be performed according to the investigator's usual routine, including pre-operative care, surgical procedure, and post-operative care, although anti-VEGF may not be given post-operatively unless there is recurrent hemorrhage.
  Interventions: Procedure: Prompt Vitrectomy Plus Panretinal Photocoagulation

INTERVENTIONS:
Drug: 2-mg Intravitreous Aflibercept Injection — Soluble decoy receptor fusion protein that has a high binding affinity to all isoforms of VEGF as well as to placental growth factor.
  Other Names: Eylea; Vascular endothelial growth factor Trap-Eye
  Arms: Intravitreous 2 mg aflibercept injections
Procedure: Prompt Vitrectomy Plus Panretinal Photocoagulation — Surgical removal of the vitreous gel and associated hemorrhage, concurrent delivery of panretinal endolaser
  Other Names: PRP
  Arms: Prompt vitrectomy plus panretinal photocoagulation

SUMMARY:
Although vitreous hemorrhage (VH) from proliferative diabetic retinopathy (PDR) can cause acute and dramatic vision loss for patients with diabetes, there is no current, evidence-based clinical guidance as to what treatment method is most likely to provide the best visual outcomes once intervention is desired. Intravitreous anti-vascular endothelial growth factor (anti-VEGF) therapy alone or vitrectomy combined with intraoperative PRP each provide the opportunity to stabilize or regress retinal neovascularization. However, clinical trials are lacking to elucidate the relative time frame of visual recovery or final visual outcome in prompt vitrectomy compared with initial anti-VEGF treatment. The Diabetic Retinopathy Clinical Research Network Protocol N demonstrated short-term trends consistent with a possible beneficial effect of anti-VEGF treatment in eyes with VH from PDR, including greater visual acuity improvement and reduced rates of recurrent VH as compared with saline injection. It is possible that a study with a longer duration of follow-up with structured anti-VEGF retreatment would demonstrate even greater effectiveness of anti-VEGF for VH to avoid vitrectomy and its attendant adverse events while also improving visual acuity. On the other hand, advances in surgical techniques leading to faster operative times, quicker patient recovery, and reduced complication rates may make prompt vitrectomy a more attractive alternative since it results in the immediate ability to clear hemorrhage and to perform PRP if desired, often as part of one procedure. This proposed study will evaluate the safety and efficacy of two treatment approaches for eyes with VH from PDR: prompt vitrectomy + PRP and intravitreous aflibercept injections.

DETAILED DESCRIPTION:
A participant could have only one eye enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years Participants <18 years old are not being included because proliferative diabetic retinopathy is so rare in this age group that the diagnosis may be questionable.
2. Diagnosis of diabetes mellitus (type 1 or type 2)

Any one of the following will be considered to be sufficient evidence that diabetes is present:

* Current regular use of insulin for the treatment of diabetes
* Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes
* Documented diabetes by American Diabetes Association and/or World Health Organization criteria 4. Able and willing to provide informed consent. 5. Patient is willing and able to undergo vitrectomy within next 2 weeks and the vitrectomy can be scheduled within that time frame.

  6. Vitreous hemorrhage causing vision impairment, presumed to be from proliferative diabetic retinopathy, for which intervention is deemed necessary.
  * Note: Prior panretinal photocoagulation is neither a requirement nor an exclusion.
  * Subhyaloid hemorrhage alone does not make an eye eligible; however, presence of subhyaloid hemorrhage in addition to the criteria above will not preclude participation provided the investigator is comfortable with either treatment regimen.

    7. Immediate vitrectomy not required (investigator and participant are willing to wait at least 4 months to see if hemorrhage clears sufficiently with anti-vascular endothelial growth factor without having to proceed to vitrectomy).

    8. Visual acuity letter score ≤78 (approximate Snellen equivalent 20/32) and at least light perception.

    9. Investigators should use particular caution when considering enrollment of an eye with visual acuity letter score 69 to 78 (approximate Snellen equivalent 20/32 to 20/40) to ensure that the need for vitrectomy and its potential benefits outweigh the potential risks.

Exclusion Criteria:

* A potential participant is not eligible if any of the following exclusion criteria are present:

  1. History of chronic renal failure requiring dialysis (including placement of fistula if performed in preparation for dialysis) or kidney transplant.
  2. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
  3. Initiation of intensive insulin treatment (a pump or multiple daily injections) within 4 months prior to randomization or plans to do so in the next 4 months.
  4. A condition that, in the opinion of the investigator, would preclude participant undergoing elective vitrectomy surgery if indicated during the study.
  5. Participation in an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval for the indication being studied.

     • Note: participants cannot receive another investigational drug while participating in the study.
  6. Known allergy to any component of the study drug or any drug used in the injection prep (including povidone iodine).
  7. Blood pressure > 180/110 (systolic above 180 or diastolic above 110).
  8. If blood pressure is brought below 180/110 by anti-hypertensive treatment, potential participant can become eligible.
  9. Systemic anti-vascular endothelial growth factor or pro-vascular endothelial growth factor treatment within 4 months prior to randomization.

     • These drugs cannot be used during the study.
  10. For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next two years.

      • Women who are potential participants should be questioned about the potential for pregnancy. Investigator judgment is used to determine when a pregnancy test is needed.
  11. Potential participant is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the two years.
  12. Evidence of traction detachment involving or threatening the macula.

      • If the density of the hemorrhage precludes a visual assessment on clinical exam to confirm eligibility, then it is recommended that assessment be performed with ultrasound as standard care.
  13. Evidence of rhegmatogenous retinal detachment.

      • If the density of the hemorrhage precludes a visual assessment on clinical exam to confirm eligibility, then it is recommended that assessment be performed with ultrasound as standard care.
  14. Evidence of neovascular glaucoma (iris or angle neovascularization is not an exclusion).
  15. Known diabetic macular edema (DME), defined as either
  16. Optical coherence tomography central subfield thickness (microns):
  17. Zeiss Cirrus: ≥290 in women; ≥305 in men
  18. Heidelberg Spectralis: ≥305 in women; ≥320 in men OR
  19. Diabetic macular edema on clinical exam that the investigator believes currently requires treatment.
  20. History of intravitreous anti-vascular endothelial growth factor treatment within 2 months prior to current vitreous hemorrhage onset or after onset.
  21. History of intraocular corticosteroid treatment within 4 months prior to current vitreous hemorrhage onset or after onset.
  22. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months or major ocular surgery other than vitrectomy anticipated within the next 6 months following randomization.
  23. History of vitrectomy.
  24. History of YAG capsulotomy performed within 2 months prior to randomization.
  25. Aphakia.
  26. Uncontrolled glaucoma (in investigator's judgment).
  27. Exam evidence of severe external ocular infection, including conjunctivitis, chalazion, or substantial blepharitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Antoszyk, MD, Study Chair — Charlotte Eye, Ear, Nose and Throat Assoc., PA
Locations (62):
- United States (60):
  - Retinal Diagnostic Center, Campbell, California
  - Macula & Retina Institute, Glendale, California
  - Atlantis Eye Care, Huntington Beach, California
  - Loma Linda University Health Care, Department of Ophthalmology, Loma Linda, California
  - Shashi D Ganti, MD PC, Porterville, California
  - Florida Retina Consultants, Lakeland, Florida
  - Southeast Eye Institute, P.A. dba Eye Associates of Pinellas, Pinellas Park, Florida
  - Retina Associates of Sarasota, Sarasota, Florida
  - Retina Associates of Florida, P.A., Tampa, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Marietta Eye Clinic, Marietta, Georgia
  - Thomas Eye Group, Sandy Springs, Georgia
  - Gailey Eye Clinic, Bloomington, Illinois
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - University of Illinois at Chicago Medical Center, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Raj K. Maturi, MD, PC, Indianapolis, Indiana
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Retina Associates, P.A., Shawnee Mission, Kansas
  - Paducah Retinal Center, Paducah, Kentucky
  - Eye Associates of Northeast Louisiana dba Haik Humble Eye Center, West Monroe, Louisiana
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Wilmer Eye Institute at Johns Hopkins, Baltimore, Maryland
  - Valley Eye Physicians and Surgeons, Ayer, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Kellogg Eye Center, University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Dept of Ophthalmology and Eye Care Services, Detroit, Michigan
  - Retina Specialists of Michigan, Grand Rapids, Michigan
  - Retina Center, PA, Minneapolis, Minnesota
  - Mayo Clinic Department of Ophthalmology, Rochester, Minnesota
  - Mid-America Retina Consultants, P.A., Kansas City, Missouri
  - The Retina Institute, St Louis, Missouri
  - The New York Eye and Ear Infirmary/Faculty Eye Practice, New York, New York
  - MaculaCare, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Retina-Vitreous Surgeons of Central New York, PC, Syracuse, New York
  - Kittner Eye Center, Chapel Hill, North Carolina
  - Charlotte Eye, Ear, Nose and Throat Assoc., PA, Charlotte, North Carolina
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Oregon Retina, LLP, Eugene, Oregon
  - Retina Northwest, PC, Portland, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Retina Vitreous Consultants, Monroeville, Pennsylvania
  - Palmetto Retina Center, West Columbia, South Carolina
  - Southeastern Retina Associates, Chattanooga, Tennessee
  - Southeastern Retina Associates, P.C., Knoxville, Tennessee
  - Southwest Retina Specialists, Amarillo, Texas
  - Retina Research Center, Austin, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Baylor Eye Physicians and Surgeons, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Valley Retina Institute, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Spokane Eye Clinic, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - UBC/VCHA Eye Care Centre, Vancouver, British Columbia
  - University Health Network - Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Beaulieu WT, Maguire MG, Antoszyk AN; DRCR Retina Network. Changes in activity impairment and work productivity after treatment for vitreous hemorrhage due to proliferative diabetic retinopathy: Secondary outcomes from a randomized controlled trial (DRCR Retina Network Protocol AB). PLoS One. 2023 Nov 16;18(11):e0293543. doi: 10.1371/journal.pone.0293543. eCollection 2023. PMID 37972038
- [Derived] Glassman AR, Beaulieu WT, Maguire MG, Antoszyk AN, Chow CC, Elman MJ, Jampol LM, Salehi-Had H, Sun JK; DRCR Retina Network. Visual Acuity, Vitreous Hemorrhage, and Other Ocular Outcomes After Vitrectomy vs Aflibercept for Vitreous Hemorrhage Due to Diabetic Retinopathy: A Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2021 Jul 1;139(7):725-733. doi: 10.1001/jamaophthalmol.2021.1110. PMID 33956075
- [Derived] Antoszyk AN, Glassman AR, Beaulieu WT, Jampol LM, Jhaveri CD, Punjabi OS, Salehi-Had H, Wells JA 3rd, Maguire MG, Stockdale CR, Martin DF, Sun JK; DRCR Retina Network. Effect of Intravitreous Aflibercept vs Vitrectomy With Panretinal Photocoagulation on Visual Acuity in Patients With Vitreous Hemorrhage From Proliferative Diabetic Retinopathy: A Randomized Clinical Trial. JAMA. 2020 Dec 15;324(23):2383-2395. doi: 10.1001/jama.2020.23027. PMID 33320223

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravitreous 2 mg Aflibercept Injections: Initial injection must be given on the day of randomization. Follow-up injections will be performed as often as every 4 weeks unless criteria for deferral are met.
  2 mg Intravitreous Aflibercept Injection: Soluble decoy receptor fusion protein that has a high binding affinity to all isoforms of vascular endothelial growth factor (VEGF) as well as to placental growth factor.
- Vitrectomy With Panretinal Photocoagulation: For the prompt vitrectomy with panretinal photocoagulation group, the vitrectomy must be scheduled to be performed within 2 weeks of randomization. Vitrectomy will be performed according to the investigator's usual routine, including pre-operative care, surgical procedure, and post-operative care, although anti-VEGF may not be given post-operatively unless there is recurrent hemorrhage.
  Vitrectomy with Panretinal Photocoagulation: Surgical removal of the vitreous gel and associated hemorrhage, concurrent delivery of panretinal endolaser
Period: Overall Study
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Vitrectomy With Panretinal Photocoagulation
Started | 100 | 105
Completed | 90 | 87
Not Completed | 10 | 18
Not completed — Death | 6 | 3
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Lost to Follow-up | 2 | 7
Not completed — Completed Out of Window | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation | Total
Number analyzed (Participants) | 100 | 105 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (12) | 57 (11) | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 43 | 90
  Male | 53 | 62 | 115
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 41 | 84
  Non-Hispanic White | 36 | 47 | 83
  Non-Hispanic Black/African American | 16 | 11 | 27
  Asian | 2 | 5 | 7
  American Indian/Alaska Native | 1 | 0 | 1
  More than one race | 1 | 0 | 1
  Unknown or not reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 100 | 105 | 205
Diabetes Type [Count of Participants; unit: Participants]
  Type 1 | 17 | 19 | 36
  Type 2 | 83 | 86 | 169
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 19 (10) | 21 (11) | 20 (11)
Insulin Used [Count of Participants; unit: Participants]
  Yes | 78 | 78 | 156
  No | 22 | 27 | 49
Hemoglobin A1c [Mean (Standard Deviation); unit: Hemoglobin A1c percentage] — Population: Hemoglobin A1c was missing for 4 and 1 eye(s) in the Intravitreous 2 mg aflibercept injections and Prompt vitrectomy plus panretinal photocoagulation groups, respectively.
  Hemoglobin A1c percentage
    number analyzed (Participants) | 96 | 104 | 200
    (all) | 8.7 (2.2) | 8.3 (1.9) | 8.5 (2.0)
Mean Arterial Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 102 (12) | 102 (12) | 102 (12)
Prior Myocardial Infarction [Count of Participants; unit: Participants] | 7 | 15 | 22
Prior Stroke [Count of Participants; unit: Participants] | 5 | 8 | 13
Kidney Disease [Count of Participants; unit: Participants] | 20 | 18 | 38
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: 15 and 12 were missing for the Aflibercept and Sham groups, respectively.
  kg/m^2
    number analyzed (Participants) | 85 | 93 | 178
    (all) | 31 (7) | 32 (7) | 31 (7)
Daily Cigarette Smoking [Count of Participants; unit: Participants]
  Never | 60 | 72 | 132
  Prior | 27 | 25 | 52
  Current | 13 | 8 | 21
Prior Treatment for Diabetic Macular Edema [Number; unit: Eyes] | 29 | 37 | 66
Prior anti-vascular endothelial growth factor for diabetic macular edema [Number; unit: Eyes] | 23 | 28 | 51
Prior anti-vascular endothelial growth factor for diabetic retinopathy [Number; unit: Eyes] | 23 | 22 | 45
Prior panretinal photocoagulation [Number; unit: Eyes] | 42 | 58 | 100
Approximate Duration of Vitreous Hemorrhage [Number; unit: Eyes]
  Less than 1 Month | 60 | 57 | 117
  1 to 3 Months | 27 | 27 | 54
  4 to 6 Months | 8 | 6 | 14
  7 to 12 Months | 1 | 6 | 7
  More than 12 Months | 4 | 9 | 13
Lens Status on Clinical Exam [Number; unit: Eyes]
  Phakic (natural lens) | 75 | 81 | 156
  Prosthetic intraocular lens | 25 | 24 | 49
E-ETDRS visual acuity letter score [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Best-corrected visual acuity following protocol-defined refraction. Visual Acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/10) to 0 letters (Snellen equivalent <20/800). Higher scores indicate better visual acuity and lower scores indicate worse visual acuity.
  units on a scale | 35.6 (28.1) | 33.5 (28.8) | 34.5 (28.4)
Traction Retinal Detachment, Macula Not Threatened [Number; unit: Eyes] | 5 | 3 | 8
Intraocular Pressure [Mean (Standard Deviation); unit: mmHg] | 16 (4) | 15 (3) | 15 (4)
Prior focal/grid laser for Diabetic Macular Edema [Number; unit: Eyes] | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: E-ETDRS Visual Acuity Letter Score (Area Under the Curve From Baseline)
Description: The area under the curve (units = letters·weeks) was divided by 24 weeks (units = weeks) to obtain an average change in letter score (units = letters) over the 24-weekr follow-up.
  Best-corrected visual acuity following protocol-defined refraction. Visual Acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/10) to 0 letters (Snellen equivalent of <20/800). Higher scores indicate better visual acuity and lower scores indicate worse visual acuity.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
Number analyzed (Participants) | 97 | 98
units on a scale | 59.3 (21.9) | 63.0 (21.7)

2. Secondary Outcome: E-ETDRS Visual Acuity Letter Score
Description: Best-corrected visual acuity following protocol-defined refraction. Visual Acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/10) to 0 letters (Snellen equivalent <20/800). Higher scores indicate better visual acuity and lower scores indicate worse visual acuity.
Time Frame: 4 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Vitrectomy With Panretinal Photocoagulation
Number analyzed (Participants) | 95 | 99
units on a scale | 52.6 (29.4) | 62.3 (26.8)

3. Secondary Outcome: E-ETDRS Visual Acuity Letter Score
Description: as for outcome 2
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
Number analyzed (Participants) | 97 | 102
units on a scale | 63.7 (25.0) | 67.3 (24.7)

4. Secondary Outcome: E-ETDRS Visual Acuity Letter Score
Description: as for outcome 2
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
Number analyzed (Participants) | 97 | 98
units on a scale | 69.4 (23.8) | 69.0 (23.1)

5. Secondary Outcome: E-ETDRS Visual Acuity Letter Score
Description: as for outcome 2
Time Frame: 1-Year from participant randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
Number analyzed (Participants) | 95 | 98
units on a scale | 70.5 (20.3) | 72.7 (20.3)

6. Secondary Outcome: E-ETDRS Visual Acuity Letter Score
Description: as for outcome 2
Time Frame: 2 Years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
Number analyzed (Participants) | 90 | 87
units on a scale | 73.7 (16.4) | 71.0 (24.0)

7. Secondary Outcome: E-ETDRS Visual Acuity Letter Score (Area Under the Curve From Baseline)
Description: Best-corrected visual acuity following protocol-defined refraction. Visual Acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/10) to 0 letters (Snellen equivalent <20/800). Higher scores indicate better visual acuity and lower scores indicate worse visual acuity. The area under the curve (units = letters·years) was divided by 2 years (units = years) to obtain an average change in letter score (units = letters) over the 2-year follow-up.
  Best-corrected visual acuity following protocol-defined refraction. Visual Acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/10) to 0 letters (Snellen equivalent of <20/800). Higher scores indicate better visual acuity and lower scores indicate worse visual acuity.
Time Frame: 2-Years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
Number analyzed (Participants) | 90 | 87
units on a scale | 68.7 (15.0) | 70.0 (18.8)

8. Secondary Outcome: Snellen Equivalent Range (Visual Acuity Score)
Description: as for outcome 2
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
Number analyzed (Participants) | 95 | 99
Participants
  20/32 or better (>=74) | 24 | 49
  20/200 or worse (<=38) | 26 | 18

9. Secondary Outcome: Snellen Equivalent Range (Visual Acuity Score)
Description: as for outcome 2
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
Number analyzed (Participants) | 97 | 102
Participants
  20/32 or better (>=74 | 45 | 58
  20/200 or worse (<=38) | 16 | 12

10. Secondary Outcome: Snellen Equivalent Range (Visual Acuity Score)
Description: as for outcome 2
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
Number analyzed (Participants) | 97 | 98
Participants
  20/32 or better (>=74 | 61 | 59
  20/200 or worse (<=38) | 10 | 10

11. Secondary Outcome: Snellen Equivalent Range (Visual Acuity Score)
Description: as for outcome 2
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
Number analyzed (Participants) | 95 | 98
Participants
  20/32 or better (>=74 | 55 | 65
  20/200 or worse (<=38) | 8 | 8

12. Secondary Outcome: Snellen Equivalent Range (Visual Acuity Score)
Description: as for outcome 2
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
Number analyzed (Participants) | 90 | 87
Participants
  20/32 or better (>=74 | 56 | 59
  20/200 or worse (<=38) | 3 | 10

13. Secondary Outcome: Recurrent Vitreous Hemorrhage
Description: Assessed by the investigator and defined as presence of vitreous hemorrhage after a period of absence. Excludes eyes in which vitreous hemorrhage could not be assessed during follow-up.
Time Frame: At any time through 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
Number analyzed (Participants) | 97 | 104
Participants | 48 | 16

14. Secondary Outcome: Retinal Neovascularization on Clinical Exam
Description: Defined as neovascularization of the disc or elsewhere. Excludes eyes in which retinal neovascularization could not be determined.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
Number analyzed (Participants) | 85 | 92
Participants | 25 | 3

15. Secondary Outcome: Retinal Neovascularization on Clinical Exam
Description: as for outcome 14
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
Number analyzed (Participants) | 89 | 95
Participants | 15 | 2

16. Secondary Outcome: Retinal Neovascularization on Clinical Exam
Description: as for outcome 14
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
Number analyzed (Participants) | 88 | 83
Participants | 20 | 2

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Intravitreous 2 mg Aflibercept Injections | Prompt Vitrectomy Plus Panretinal Photocoagulation
All-Cause Mortality (participants affected / at risk) | 6/100 | 3/105
Serious Adverse Events (participants affected / at risk) | 44/100 | 45/105
Other Adverse Events (participants affected / at risk) | 97/100 | 98/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravitreous 2 mg Aflibercept Injections (N=100) | Prompt Vitrectomy Plus Panretinal Photocoagulation (N=105)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphangitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Bicuspid aortic valve (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (3) | 0 (0)
Congestive heart failure (Cardiac disorders) | 4 (6) | 4 (5)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Heart failure (Cardiac disorders) | 1 (1) | 2 (2)
Mitral valve disorders (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Unstable angina (Cardiac disorders) | 1 (1) | 0 (0)
Diabetes (Endocrine disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Endocrine disorders) | 4 (7) | 2 (3)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Hyperglycemic hyperosmolar nonketotic syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Hypoglycemia (Endocrine disorders) | 1 (1) | 1 (1)
Loss of control of blood sugar (Endocrine disorders) | 0 (0) | 1 (1)
Endophthalmitis (Eye disorders) | 1 (1) | 2 (2)
Exposure keratoconjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Ischemia retinal (Eye disorders) | 0 (0) | 1 (1)
Ocular fundus arteriosclerosis (Eye disorders) | 0 (0) | 1 (1)
Rhegmatogenous retinal detachment (Eye disorders) | 2 (3) | 0 (0)
Traction retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Visual acuity decreased (Eye disorders) | 1 (1) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (4) | 0 (0)
Hyperemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Leg edema (General disorders) | 1 (1) | 1 (1)
Peripheral edema (General disorders) | 1 (1) | 0 (0)
Acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Abscess NOS (Infections and infestations) | 0 (0) | 2 (2)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Foot infection (Infections and infestations) | 6 (6) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
MRSA (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 5 (6) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heart rate low (Investigations) | 0 (0) | 2 (2)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fluid overload - fluid volume increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type II diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Water retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Broken bones (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Femur fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fractured collar bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fractured ribs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hip fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0)
Pulled hamstring (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Viral meningitis (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (3)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic renal failure worsened (Renal and urinary disorders) | 0 (0) | 1 (2)
End stage renal disease (ESRD) (Renal and urinary disorders) | 1 (1) | 1 (1)
Kidney failure (Renal and urinary disorders) | 7 (7) | 1 (2)
Kidney infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Kidney stones (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Testicular torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Cardiopulmonary arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Cellulitis of arm (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Cellulitis of foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cellulitis of leg (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cellulitis of toe (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic foot ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Foot ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Back surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Bypass surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary artery bypass graft (Surgical and medical procedures) | 1 (1) | 0 (0)
Foot surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee surgery NOS (Surgical and medical procedures) | 0 (0) | 1 (1)
Metatarsal excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Stent placement (Surgical and medical procedures) | 0 (0) | 2 (2)
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Embolism - blood clot (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypertension worsened (Vascular disorders) | 3 (4) | 2 (2)
Hypotension (Vascular disorders) | 2 (3) | 1 (1)
Intraventricular hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Ischemia - systemic (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disease (Vascular disorders) | 1 (1) | 0 (0)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
Stroke (cerebrovascular accident) (Vascular disorders) | 0 (0) | 1 (1)
Stroke - Ischemic (Vascular disorders) | 1 (1) | 0 (0)
Transient ischemic attacks (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravitreous 2 mg Aflibercept Injections (N=100) | Prompt Vitrectomy Plus Panretinal Photocoagulation (N=105)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 7 (8)
Anemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anemia, unspecified (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arteriosclerotic heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1)
Congestive heart failure (Cardiac disorders) | 2 (2) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0)
Ischemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial disorder (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary valve regurgitation (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid regurgitation (Cardiac disorders) | 1 (1) | 0 (0)
Anomaly heart (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear infection (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Otitis media acute (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diabetes (Endocrine disorders) | 1 (1) | 1 (1)
Diabetes mellitus poor control (Endocrine disorders) | 1 (1) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1) | 2 (2)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypoglycemia (Endocrine disorders) | 5 (6) | 3 (3)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Loss of control of blood sugar (Endocrine disorders) | 1 (1) | 3 (3)
Worsening of diabetes (Endocrine disorders) | 3 (3) | 2 (2)
Allergic conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Anterior chamber angle neovascularisation (Eye disorders) | 3 (3) | 1 (1)
Anterior chamber cell (Eye disorders) | 4 (4) | 3 (4)
Anterior chamber flare (Eye disorders) | 2 (2) | 2 (2)
Atrophy of macula (Eye disorders) | 0 (0) | 1 (1)
Band keratopathy (Eye disorders) | 0 (0) | 1 (1)
Blepharitis (eyelid irritation) (Eye disorders) | 1 (1) | 2 (2)
Blurred vision (Eye disorders) | 9 (10) | 3 (3)
Blurry vision (Eye disorders) | 10 (11) | 3 (3)
Cataract (Eye disorders) | 14 (14) | 20 (23)
Cataract cortical (Eye disorders) | 5 (5) | 1 (2)
Cataract fragments in eye postoperative (Eye disorders) | 0 (0) | 1 (1)
Cataract subcapsular (Eye disorders) | 1 (1) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 1 (1)
Choroidal detachment (Eye disorders) | 0 (0) | 2 (2)
Cloudy vision (Eye disorders) | 0 (0) | 4 (4)
Conjunctival cyst (Eye disorders) | 0 (0) | 1 (1)
Conjunctival hyperemia (Eye disorders) | 0 (0) | 1 (2)
Corneal abrasion (Eye disorders) | 3 (3) | 2 (2)
Corneal defect (Eye disorders) | 1 (1) | 1 (1)
Corneal disorder (NOS) (Eye disorders) | 0 (0) | 1 (1)
Corneal edema (Eye disorders) | 0 (0) | 5 (5)
Corneal endothelial disorder (Eye disorders) | 1 (1) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 1 (1)
Corneal guttata (Eye disorders) | 0 (0) | 1 (1)
Corneal haze (Eye disorders) | 0 (0) | 1 (1)
Corneal irritation (Eye disorders) | 0 (0) | 2 (2)
Corneal scar (Eye disorders) | 0 (0) | 1 (1)
Corneal ulcer (Eye disorders) | 0 (0) | 2 (2)
Cortical spoking (Eye disorders) | 7 (7) | 2 (2)
Cupping of optic nerve (Eye disorders) | 0 (0) | 1 (1)
Decrease in depth perception (Eye disorders) | 1 (1) | 0 (0)
Detachment of retinal pigment epithelium (Eye disorders) | 0 (0) | 1 (1)
Diabetic macular edema (Eye disorders) | 10 (11) | 9 (11)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Disc neovascularization (Eye disorders) | 7 (7) | 0 (0)
Double vision (Eye disorders) | 2 (2) | 2 (2)
Dry eye (Eye disorders) | 6 (6) | 7 (7)
Dry eye syndrome (Eye disorders) | 1 (1) | 1 (1)
Epiretinal membrane (Eye disorders) | 12 (13) | 13 (13)
Exposure keratoconjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Eye ache (Eye disorders) | 1 (1) | 1 (1)
Eye irritation (Eye disorders) | 2 (2) | 5 (5)
Eye itching (Eye disorders) | 3 (5) | 7 (7)
Eye pain (Eye disorders) | 11 (14) | 6 (7)
Eye strain (Eye disorders) | 1 (1) | 0 (0)
Eye tearing (Eye disorders) | 2 (2) | 1 (1)
Eyelid edema (Eye disorders) | 0 (0) | 1 (1)
Eyelid pain (Eye disorders) | 1 (1) | 0 (0)
Eyelid twitching (Eye disorders) | 0 (0) | 1 (1)
Filmy vision (Eye disorders) | 1 (1) | 0 (0)
Flame-shaped hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 24 (30) | 11 (11)
Folds in Descemet's membrane (Eye disorders) | 0 (0) | 1 (1)
Foreign body in conjunctival sac (Eye disorders) | 0 (0) | 2 (2)
Foreign body sensation in eyes (Eye disorders) | 2 (2) | 4 (4)
Glare (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 2 (2) | 4 (5)
Hazy vision (Eye disorders) | 4 (4) | 1 (1)
Hordeolum (Eye disorders) | 1 (1) | 0 (0)
Hypertensive retinopathy (Eye disorders) | 1 (1) | 1 (1)
Hyphema (Eye disorders) | 0 (0) | 4 (5)
Hypotony of eye (Eye disorders) | 0 (0) | 1 (1)
Intraretinal microvascular abnormalities (Eye disorders) | 2 (4) | 0 (0)
Iris neovascularization (Eye disorders) | 2 (2) | 2 (2)
Iritis (anterior uveitis, iridocyclitis) (Eye disorders) | 1 (2) | 1 (1)
Ischemia retinal (Eye disorders) | 0 (0) | 1 (1)
Keratopathy NOS (Eye disorders) | 0 (0) | 1 (1)
Lattice degeneration of retina (Eye disorders) | 1 (1) | 0 (0)
Macular atrophy (Eye disorders) | 1 (1) | 0 (0)
Macular dystrophy (Eye disorders) | 0 (0) | 1 (1)
Macular edema (Eye disorders) | 0 (0) | 1 (1)
Macular hole (Eye disorders) | 2 (2) | 0 (0)
Macular puckering (Eye disorders) | 1 (1) | 2 (2)
Macular scar (Eye disorders) | 0 (0) | 1 (1)
Meibomian gland obstruction (Eye disorders) | 0 (0) | 1 (1)
Neovascular glaucoma (Eye disorders) | 1 (1) | 2 (2)
Neurosensory detachment (Eye disorders) | 0 (0) | 1 (1)
Nuclear sclerosis (Eye disorders) | 15 (16) | 10 (10)
Ocular discomfort (Eye disorders) | 2 (2) | 0 (0)
Ocular hypertension (Eye disorders) | 3 (3) | 3 (3)
Optic nerve pallor (Eye disorders) | 2 (2) | 0 (0)
Photophobia (Eye disorders) | 3 (3) | 1 (1)
Photopsia (Eye disorders) | 1 (1) | 1 (1)
Posterior capsule opacification (Eye disorders) | 10 (11) | 11 (12)
Posterior subcapsular cataract (Eye disorders) | 16 (19) | 16 (19)
Posterior vitreous detachment (Eye disorders) | 2 (2) | 0 (0)
Preretinal fibrosis (Eye disorders) | 2 (2) | 0 (0)
Preretinal hemorrhage (Eye disorders) | 3 (3) | 0 (0)
Proliferative vitreoretinopathy (Eye disorders) | 1 (1) | 0 (0)
Ptosis (Eye disorders) | 0 (0) | 2 (2)
Punctate epithelial erosion (Eye disorders) | 3 (3) | 0 (0)
Red eye (Eye disorders) | 1 (2) | 0 (0)
Retinal cyst (Eye disorders) | 0 (0) | 1 (1)
Retinal edema (Eye disorders) | 1 (1) | 2 (2)
Retinal exudates (Eye disorders) | 4 (5) | 3 (3)
Retinal hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Retinal macroaneurysm (Eye disorders) | 1 (1) | 0 (0)
Retinal neovascularization (Eye disorders) | 7 (9) | 3 (3)
Retinal tear (Eye disorders) | 7 (7) | 5 (5)
Retinal vessel avulsion (Eye disorders) | 2 (2) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 2 (2) | 2 (2)
Rubeosis iridis (Eye disorders) | 0 (0) | 3 (3)
Secondary cataract (Eye disorders) | 1 (1) | 0 (0)
Senile nuclear sclerosis (Eye disorders) | 0 (0) | 1 (1)
Sensation of pressure in eye (Eye disorders) | 0 (0) | 1 (1)
Sensitivity to light (photophobia) (Eye disorders) | 2 (2) | 4 (4)
Soreness in eyes (Eye disorders) | 3 (5) | 0 (0)
Stye (Eye disorders) | 0 (0) | 1 (1)
Subconjunctival hemorrhage (Eye disorders) | 3 (3) | 4 (4)
Subconjunctival/conjunctival hemorrhage (Eye disorders) | 0 (0) | 1 (1)
Subretinal fibrosis (Eye disorders) | 0 (0) | 1 (1)
Subretinal hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Superficial punctate keratitis (Eye disorders) | 3 (3) | 2 (2)
Swollen eyelid (Eye disorders) | 1 (1) | 0 (0)
Swollen eyes (Eye disorders) | 2 (2) | 0 (0)
Synechiae (Eye disorders) | 1 (1) | 0 (0)
Traction retinal detachment (Eye disorders) | 20 (23) | 2 (3)
Varying retinal vessel calibre (Eye disorders) | 1 (1) | 0 (0)
Vision decreased (Eye disorders) | 11 (11) | 5 (6)
Vision peripheral decreased (Eye disorders) | 0 (0) | 1 (1)
Visual acuity decreased (Eye disorders) | 3 (4) | 1 (1)
Visual disturbances (Eye disorders) | 2 (2) | 1 (1)
Visual flashes (Eye disorders) | 3 (5) | 5 (5)
Vitreoretinal traction syndrome (Eye disorders) | 1 (1) | 0 (0)
Vitreous debris (Eye disorders) | 3 (3) | 0 (0)
Vitreous disorder NOS (Eye disorders) | 1 (1) | 0 (0)
Vitreous floater (Eye disorders) | 2 (2) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 52 (75) | 24 (31)
Vitreous membranes and strands (Eye disorders) | 0 (0) | 1 (1)
Vitreous opacities (Eye disorders) | 1 (1) | 0 (0)
Vitreous opacity (Eye disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (4)
Acid reflux (oesophageal) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Barrett's esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloody stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chipped tooth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 6 (8) | 1 (1)
Distention (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
External hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroesophageal reflux (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 7 (7)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Stomach virus (Gastrointestinal disorders) | 2 (2) | 2 (2)
Tooth abscess (Gastrointestinal disorders) | 1 (3) | 0 (0)
Tooth infection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upset stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (8) | 2 (2)
Anasarca (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 4 (4) | 1 (1)
Chronic pain (General disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 1 (1) | 1 (1)
Dialysis access malfunction (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 2 (2)
General Swelling (General disorders) | 1 (1) | 1 (1)
Leg edema (General disorders) | 4 (4) | 1 (1)
Localized superficial swelling, mass, or lump (General disorders) | 0 (0) | 1 (1)
Pain NOS (General disorders) | 0 (0) | 1 (1)
Pedal edema (General disorders) | 1 (1) | 0 (0)
Swelling of feet (General disorders) | 2 (2) | 1 (1)
Acute cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallstones (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatopathy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver enlargement (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (2) | 0 (0)
Hives (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 3 (3) | 1 (1)
Specific allergy (drug) (Immune system disorders) | 0 (0) | 1 (1)
Abscess NOS (Infections and infestations) | 0 (0) | 1 (1)
Acute pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Foot infection (Infections and infestations) | 1 (1) | 2 (2)
Fungal infection of nail (Infections and infestations) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 2 (2)
Gum infection (Infections and infestations) | 1 (1) | 0 (0)
Infected toe (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (3)
Influenza (Infections and infestations) | 10 (10) | 10 (10)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
MRSA (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Streptococcal infection NOS (Infections and infestations) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 1 (1) | 0 (0)
Viral syndrome (Infections and infestations) | 0 (0) | 1 (1)
Yeast infection (Infections and infestations) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bee sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Black eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bug bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 8 (9) | 3 (3)
Foot injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Knee injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Laceration of leg (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Phlebitis - Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Blood sugar decreased (Investigations) | 1 (1) | 1 (1)
Hormonal imbalance (Investigations) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 7 (7) | 9 (10)
Laboratory test abnormal (Investigations) | 1 (1) | 1 (2)
Oxygen saturation low (Investigations) | 0 (0) | 1 (1)
Potassium high (Investigations) | 0 (0) | 1 (1)
Abnormal weight gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Fluid overload - fluid volume increased (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypercholesterolemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Magnesium deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Morbid obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B6 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Water retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis NOS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Back strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone spur (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Broken bones (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Broken foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Charcot arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Degenerative disc disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dislocated shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Fractured ribs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Frozen shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Hand pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hip fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc bulging (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Muscle pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Sprained ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sprains and strains of ribs (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Wrist fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Wrist pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Concussion (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Head pain (Nervous system disorders) | 2 (2) | 0 (0)
Head pressure (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 9 (9) | 7 (7)
Migraine headache (Nervous system disorders) | 3 (4) | 0 (0)
Neuropathy (Nervous system disorders) | 4 (4) | 0 (0)
Numbness in hand (Nervous system disorders) | 0 (0) | 1 (1)
Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Restless leg syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
VIth nerve palsy (Nervous system disorders) | 0 (0) | 2 (2)
Vertigo (Nervous system disorders) | 1 (1) | 4 (4)
Deposit on the surface of intraocular lens (Product Issues) | 1 (1) | 0 (0)
Adjustment disorder NOS (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (4) | 7 (7)
Chronic renal failure worsened (Renal and urinary disorders) | 1 (1) | 2 (2)
End stage renal disease (ESRD) (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Kidney failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Kidney function abnormal (Renal and urinary disorders) | 2 (2) | 0 (0)
Kidney infection (Renal and urinary disorders) | 2 (2) | 1 (1)
Kidney stones (Renal and urinary disorders) | 3 (3) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
Uremia (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary hesitancy (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 8 (13) | 7 (9)
Enlarged prostate (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Hydrocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine fibroid (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvodynia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cold (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 7 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (4)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blister of foot and toe(s), without mention of infection (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Bruise (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Cellulitis of foot (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Cellulitis of toe (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatochalasis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Diabetic foot ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Epidermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythematous conditions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Foot ulcer (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (5)
Fungal infection of nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Mole of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Sebaceous cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin cancer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling of face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Benign tumor excision (Surgical and medical procedures) | 1 (1) | 1 (1)
Carpal tunnel release (Surgical and medical procedures) | 1 (1) | 0 (0)
Cataract extraction (Surgical and medical procedures) | 2 (2) | 1 (1)
Coronary stent placement (Surgical and medical procedures) | 0 (0) | 1 (1)
Foot surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Sinus operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin graft (Surgical and medical procedures) | 1 (18) | 0 (0)
Surgery (Surgical and medical procedures) | 2 (2) | 2 (2)
Toe amputation (Surgical and medical procedures) | 0 (0) | 3 (3)
Tooth extraction (Surgical and medical procedures) | 3 (3) | 3 (3)
Vitrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Wrist surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriovenous graft site hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Benign essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 4 (4)
Hypertension worsened (Vascular disorders) | 6 (7) | 3 (3)
Hypertensive crisis (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 1 (1)
Iliac artery blockage (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial disease (Vascular disorders) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
Venous malformation NOS (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT02858076/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT02858076/SAP_001.pdf
  • Informed Consent Form (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT02858076/ICF_002.pdf